CLINICAL TRIAL: NCT06126640
Title: A Phase III, Multicenter, Randomized, Open-Label, Active-Controlled Study of SHR-A1811 Versus Trastuzumab Emtansine (T-DM1) in HER2-Positive Primary Breast Cancer Participants With Residual Invasive Disease Following Neoadjuvant Therapy
Brief Title: A Phase III, Active-Controlled Study of SHR-A1811 Versus Trastuzumab Emtansine (T-DM1) in HER2-Positive Primary Breast Cancer Participants With Residual Invasive Disease Following Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-305
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: HER2-Positive Primary Breast Cancer Participants With Residual Invasive Disease Following Neoadjuvant Therapy
MeSH Terms: interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- Trastuzumab Emtansine (T-DM1) (Active Comparator)
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: SHR-A1811 — Lyophilized powder injection, 100mg / bottle, intravenous drip
  Arms: SHR-A1811
Drug: Trastuzumab Emtansine — Lyophilized powder injection, 160mg / bottle, 100mg / bottle, intravenous drip
  Arms: Trastuzumab Emtansine (T-DM1)

SUMMARY:
This study aims to Active-Controlled Study of SHR-A1811 Versus Trastuzumab Emtansine (T-DM1) in HER2-Positive Primary Breast Cancer Participants with Residual Invasive Disease Following Neoadjuvant Therapy，This study will examine SHR-A1811versus trastuzumab emtansine (T-DM1) in patients with HER2-positive primary breast cancer who have residual invasive disease in breast or axillary lymph nodes after neoadjuvant therapy.The primary objective is to compare invasive disease-free survival (IDFS) between SHR-A1811 and T-DM1 treatment arms in this population. The key secondary objective of the study is to evaluate disease-free survival (DFS), overall survival (OS) and distant recurrence-free interval (DRFI).

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18-75 years old (including both ends), and female
2. HER2 positive invasive breast cancer Confirmed by pathological examination
3. Clinical Stage before Neoadjuvant Therapy was T1-4, N0-3, M0 (excluding T1N0).
4. Residual invasive cancer confirmed by pathological examination after radical surgery must meet one of the following two conditions:

   * If the clinical stage before neoadjuvant therapy is cT4N0-3M0 or cT1-3N2-3M0, there is residual invasive cancer in the primary breast lesion and/or ipsilateral axillary lymph nodes after surgery.
   * If the clinical stage before neoadjuvant therapy was cT1-3N0-1M0 (except T1N0), there was residual invasive cancer in the ipsilateral axillary lymph nodes after surgery.
5. Previous neoadjuvant therapy must meet all of the following conditions:

   * Neoadjuvant chemotherapy: At least 6 treatment cycles, including no less than 9 weeks of taxane-based chemotherapy (anthracycline-containing chemotherapy allowed).
   * Neoadjuvant anti-HER2 targeted therapy: No less than 9 weeks of targeted therapy including trastuzumab must be completed.
6. Have received radical surgery for breast cancer:
7. The interval from the completion of radical surgery to the first random medication should be at least 3 weeks and no more than 12 weeks.
8. Hormone receptor (HR) status was confirmed by postoperative pathologic examination. HR positive is defined as positive for the estrogen receptor (ER) or progesterone receptor (PR), and HR negative is defined as negative for both ER and PR.
9. The ECOG score is 0 or 1
10. Heart function is good
11. Agree to birth control

Exclusion Criteria:

1. Stage IV metastatic breast cancer
2. Evidence of recurrent breast cancer, including local recurrence, regional recurrence and distant metastasis .
3. In the past 5 years, patients suffered from other malignant tumors, excluding cured basal cell carcinoma of skin andcervical carcinoma in situ,.
4. Previously received systemic anti-HER2-ADC drug therapy, including but not limited to trastuzumab emtansine (T-DM1), Trastuzumab Deruxtecan (T-DXd), etc.
5. Previous dosage requirements for anthracycline exposure meet one of the following conditions:

   * Doxorubicin or anthracyclines with similar exposure equivalent > 240mg/m2;
   * Epirubicin or liposomal doxorubicin hydrochloride > 480mg/m2.
6. History of cardiovascular diseases with clinical significance, such as severe/unstable angina pectoris, symptomatic congestive heart failure (NYHA ≥ Ⅱ), supraventricular or ventricular arrhythmia with clinical significance and requiring treatment or intervention, and myocardial infarction within 6 months.
7. Subjects with known or suspected interstitial pneumonia.
8. Known hereditary or acquired bleeding and thrombosis tendency.
9. History of active hepatitis B, hepatitis C or liver cirrhosis.
10. There were other serious physical or mental diseases or abnormal laboratory examinations that may increase the risk of participating in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | Randomization until the disease progressed, up to approximately 77 months postdose

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Randomization until the disease progressed, up to approximately 77 months postdose
Overall survival(OS) | Randomization until death from any cause, up to approximately 101 months postdose.
Distant recurrence-free interval (DRFI) | Randomization until distant recurrence or death from any cause, up to approximately 101 months postdose.
Safety endpointPercentage of Adverse Events in Participants | Baseline up to approximately 101 months postdose

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided